CLINICAL TRIAL: NCT01036932
Title: To Study the Safety and Efficacy of G-CSF Therapy on the CD 34 Cell Mobilization and Outcome of Patients With ACLF
Brief Title: Granulocyte Colony Stimulating Factor(G-CSF) Therapy for Patients With ACLF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Govind Ballabh Pant Hospital (Other Government)
Responsible Party: Dr S.K.Sarin, Head, Gastroenterology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IEC MAMC 179
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Last update posted 2009-12-21 (Estimated); Status verified 2009-12

CONDITIONS: Acute on Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — Granulocyte Colony-Stimulating Factor; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G-CSF group (Active Comparator): Patients with Acute on chronic liver failure after baseline investigations for the etiology of the acute event and the underlying chronic disease were given Granulocyte Colony Stimulating Factor therapy for a total duration of one month.
  Interventions: Drug: Granulocyte Colony Stimulating Factor
- Placebo (Placebo Comparator): After baseline characterization and work up for underlying acute and chronic liver disease, patients were given placebo along with the standard therapy
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Granulocyte Colony Stimulating Factor — Dose of 5 µg/kg s/c at days 1, 2, 3, 4, 5, and then every 3rd day till day 28 (total 12 doses) along with the standard therapy.
  Arms: G-CSF group
Drug: Normal Saline — dose of 1ml s/c at days 1, 2, 3, 4, 5, and then every 3rd day till day 28 (total 12 doses) along with the standard therapy.
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether Granulocyte Colony Stimulating factor(G-CSF) therapy is effective in the treatment of patients with Acute on chronic liver failure(ACLF). The investigators hypothesize that ACLF is a disease where severe hepatic impairment is accompanied by impaired hepatic regeneration. BMC mobilization using G-CSF therapy, or G-CSF therapy per se would increase the regenerative capacity of the liver and shall lead to clinical, biochemical and histological improvements in patients with ACLF.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute hepatic insult manifesting as jaundice (Sr. Bil. ≥5 mg/dL) and coagulopathy (INR≥1.5), complicated within 4 weeks by ascites and/or encephalopathy in a patient with previously diagnosed or undiagnosed chronic liver disease.(APASL criteria)

Exclusion Criteria:

* HCC or portal vein thrombosis. Refusal to participate in the study. Sepsis ( Any culture positive: blood, urine, focus of infection on Xray chest, any other obvious source of infection: UTI, SBP) Multi organ failure. Grade 3 or 4 hepatic encephalopathy.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
mobilization of CD34 cells in the peripheral blood | 1 month

SECONDARY OUTCOMES:
clinical/ biochemical improvement in liver function profile | 2 months
frequency of multi-organ failure | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Shiv K Sarin, MD, DM, Principal Investigator — G B Pant Hospital, New Delhi, India
Locations (1):
- Shiv K Sarin, New Delhi, New Delhi, India

REFERENCES:
- [Derived] Garg V, Garg H, Khan A, Trehanpati N, Kumar A, Sharma BC, Sakhuja P, Sarin SK. Granulocyte colony-stimulating factor mobilizes CD34(+) cells and improves survival of patients with acute-on-chronic liver failure. Gastroenterology. 2012 Mar;142(3):505-512.e1. doi: 10.1053/j.gastro.2011.11.027. Epub 2011 Nov 23. PMID 22119930